CLINICAL TRIAL: NCT01945281
Title: A Multicenter, Double-Blind, Randomized, Comparator-Controlled Study to Evaluate the Safety, Tolerability, and Efficacy of Caspofungin Versus Amphotericin B Deoxycholate in the Treatment of Invasive Candidiasis in Neonates and Infants Less Than 3 Months of Age
Brief Title: Safety, Tolerability, and Efficacy of Caspofungin Versus Amphotericin B Deoxycholate in the Treatment of Invasive Candidiasis in Neonates and Infants (MK-0991-064)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Operational feasibility with low recruitment due to changing epidemiology of disease
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0991-064; 2013-002084-26 (EudraCT Number); MK-0991-064 (Other: Merck Protocol Number)
Record Dates: First submitted 2013-09-13; First posted 2013-09-18 (Estimated); Results first posted 2018-08-28 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Candidiasis, Invasive
MeSH Terms: conditions — Candidiasis, Invasive | interventions — Caspofungin; amphotericin B, deoxycholate drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Caspofungin (Experimental): Caspofungin 2 mg/kg intravenous once daily for ≥14 days after documented negative culture and improvement of clinical signs and symptoms, for a maximum of 90 days treatment
  Interventions: Drug: Caspofungin
- Amphotericin B Deoxycholate (Active Comparator): Amphotericin B deoxycholate 1 mg/kg intravenous once daily for ≥14 days after documented negative culture and improvement of clinical signs and symptoms, for a maximum of 90 days treatment
  Interventions: Drug: Amphotericin B Deoxycholate

INTERVENTIONS:
Drug: Caspofungin
  Arms: Caspofungin
Drug: Amphotericin B Deoxycholate
  Arms: Amphotericin B Deoxycholate

SUMMARY:
The study will evaluate the safety, tolerability, and efficacy of caspofungin as compared with amphotericin B deoxycholate in the treatment of invasive candidiasis in neonates and infants. The primary hypothesis to be tested in the study is that caspofungin will be superior to amphotericin B deoxycholate with regard to the proportion of participants with fungal-free survival at the 2-week post-therapy follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Culture-confirmed invasive Candida infection

Exclusion Criteria:

* Candida disease limited to the oropharynx, esophagus, or other mucosal or superficial skin surfaces
* Positive culture for Candida only from sputum, broncho-alveolar lavage, catheter tip, or previously placed indwelling non-vascular catheters or drains
* Prosthetic device as the suspected site of Candida infection
* Active co-infection with a non-Candida fungal organism
* Received >48 hours of systemic antifungal treatment since the positive Candida index culture was collected as therapy for the present episode of invasive candidiasis
* Failed prior systemic antifungal therapy for the present episode of invasive candidiasis
* Diagnosis of acute hepatitis or cirrhosis
* Scheduled or anticipated to receive rifampin or other systemic antifungal therapy while on study therapy
* History (including participant's mother) of allergy, hypersensitivity, or any serious reaction to caspofungin or other member of the echinocandin class, or to amphotericin B deoxycholate or other member of the polyene class
* Severe congenital disorder known to lower immune response

Max Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2014-01-15 (Actual); Primary Completion 2018-01-02 (Actual); Study Completion 2018-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Kim J, Nakwa FL, Araujo Motta F, Liu H, Dorr MB, Anderson LJ, Kartsonis N. A randomized, double-blind trial investigating the efficacy of caspofungin versus amphotericin B deoxycholate in the treatment of invasive candidiasis in neonates and infants younger than 3 months of age. J Antimicrob Chemother. 2020 Jan 1;75(1):215-220. doi: 10.1093/jac/dkz398. PMID 31586424

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants less than 3 months of age with invasive candidiasis were enrolled in this study.
Period: Overall Study
Arm/Group | Caspofungin | Amphotericin B Deoxycholate
Started | 34 | 17
Treated | 33 | 16
Completed | 28 | 13
Not Completed | 6 | 4
Not completed — Adverse Event | 1 | 0
Not completed — Death | 3 | 3
Not completed — Physician Decision | 1 | 1
Not completed — Technical Problems | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Caspofungin | Amphotericin B Deoxycholate | Total
Number analyzed (Participants) | 34 | 17 | 51
Age, Continuous [Mean (Standard Deviation); unit: Days] | 31.1 (20.9) | 32.8 (23.3) | 31.7 (21.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 10 | 24
  Male | 20 | 7 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 7 | 19
  Not Hispanic or Latino | 19 | 9 | 28
  Unknown or Not Reported | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 1 | 4
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 6 | 19
  White | 13 | 8 | 21
  More than one race | 5 | 2 | 7
  Unknown or Not Reported | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: Grams] — Weight at Baseline Measurement Population: Participants who received at least 1 full dose of study therapy and had a documented (culture-confirmed) diagnosis of invasive candidiasis.
  Grams
    number analyzed (Participants) | 31 | 16 | 47
    (all) | 1982.1 (980.6) | 2160.9 (1513.8) | 2042.9 (1175.5)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Fungal-free Survival Through the 2-week Post-therapy Period
Description: Fungal-free survival is those participants who survived up to 2 weeks post-therapy, and had documented microbiological eradication of Candida species (sp.) from follow-up cultures collected after the initiation of study therapy. Microbiological eradication denotes negative follow-up cultures for Candida sp. from the site of infection. If a culture is not obtained on the day of assessment, the last culture after study entry may be used to assist in the assessment of microbiological eradication. If the last culture is negative for Candida sp., then microbiological eradication would be considered achieved.
Time Frame: Up to 104 days
Population: Participants who received at least 1 full dose of study therapy and had a documented (culture-confirmed) diagnosis of invasive candidiasis.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Caspofungin | Amphotericin B Deoxycholate
Number analyzed (Participants) | 31 | 16
Percentage of Participants | 71.0 [52.0 to 85.8] | 68.8 [41.3 to 89.0]
Statistical Analysis 1: Comparison: Caspofungin vs Amphotericin B Deoxycholate; Test type: Other — Miettinen & Nurminen method stratified by stratum (Weight category based on weight at study entry) with Cochran Mantel-Haenszel's weights; Difference in Percentage = -0.9, 95% CI 2-sided [-24.3 to 27.7] — Caspofungin minus Amphotericin

2. Secondary Outcome: Percentage of Participants With Fungal-free Survival Through the End of Study Treatment
Description: Fungal-free survival is those participants who survived up to end of study treatment, and had documented microbiological eradication of Candida sp. from follow-up cultures collected after the initiation of study therapy. Microbiological eradication denotes negative follow-up cultures for Candida sp. from the site of infection. If a culture is not obtained on the day of assessment, the last culture after study entry may be used to assist in the assessment of microbiological eradication. If the last culture is negative for Candida sp., then microbiological eradication would be considered achieved.
Time Frame: Up to 90 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Caspofungin | Amphotericin B Deoxycholate
Number analyzed (Participants) | 31 | 16
Percentage of Participants | 71.0 [52.0 to 85.8] | 75.0 [47.6 to 92.7]
Statistical Analysis 1: Comparison: Caspofungin vs Amphotericin B Deoxycholate; Test type: Other — [test comment as in outcome 1, analysis 1]; Difference in Percentage = -6.3, 95% CI 2-sided [-30.2 to 22.6] — Caspofungin minus Amphotericin

3. Secondary Outcome: Number of Participants With an Adverse Event (AE)
Description: An AE is any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the SPONSOR's product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which is temporally associated with the use of the SPONSOR's product, is also an AE.
Time Frame: 8 weeks after end of study therapy (up to 146 days)
Population: All participants as treated
Measure: Count of Participants; unit: Participants
Arm/Group | Caspofungin | Amphotericin B Deoxycholate
Number analyzed (Participants) | 33 | 16
Participants | 28 | 16

ADVERSE EVENTS:
Time Frame: 8 weeks after end of study therapy (up to 146 days)
Description: All participants as treated
Arm/Group | Caspofungin | Amphotericin B Deoxycholate
All-Cause Mortality (participants affected / at risk) | 2/33 | 3/16
Serious Adverse Events (participants affected / at risk) | 7/33 | 9/16
Other Adverse Events (participants affected / at risk) | 23/33 | 15/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Caspofungin (N=33) | Amphotericin B Deoxycholate (N=16)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Necrotising colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Necrotising enterocolitis neonatal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bacterial sepsis (Infections and infestations) | 0 (0) | 1 (1)
Bronchiolitis (Infections and infestations) | 0 (0) | 1 (1)
Device related sepsis (Infections and infestations) | 0 (0) | 1 (1)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0)
Escherichia sepsis (Infections and infestations) | 1 (1) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1)
Meningitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia escherichia (Infections and infestations) | 0 (0) | 2 (2)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Anastomotic complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural pneumothorax (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Suture rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Superior vena cava syndrome (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Caspofungin (N=33) | Amphotericin B Deoxycholate (N=16)
Anaemia (Blood and lymphatic system disorders) | 10 (16) | 8 (12)
Leukostasis syndrome (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 2 (3)
Tachycardia (Cardiac disorders) | 2 (2) | 2 (2)
Eye discharge (Eye disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (2) | 2 (2)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1)
Necrotising enterocolitis neonatal (Gastrointestinal disorders) | 1 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (4) | 1 (2)
Hypothermia (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 6 (10) | 3 (6)
Cholestasis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Jaundice (Hepatobiliary disorders) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 3 (5) | 5 (6)
Septic shock (Infections and infestations) | 1 (1) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 3 (3)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (2)
Blood bilirubin increased (Investigations) | 0 (0) | 2 (2)
Blood bilirubin unconjugated increased (Investigations) | 0 (0) | 1 (3)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (1)
Blood potassium increased (Investigations) | 2 (2) | 0 (0)
Blood triglycerides increased (Investigations) | 0 (0) | 1 (1)
Oxygen saturation decreased (Investigations) | 0 (0) | 1 (1)
Feeding intolerance (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypochloraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (3) | 2 (5)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Metabolic alkalosis (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Seizure (Nervous system disorders) | 1 (5) | 1 (1)
Glycosuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal tubular necrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The trial was terminated early due to operational feasibility with low recruitment due to changing epidemiology of disease.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-08-27): https://cdn.clinicaltrials.gov/large-docs/81/NCT01945281/Prot_SAP_000.pdf